CLINICAL TRIAL: NCT01540279
Title: Do Antibacterial Skin Sutures Reduce Surgical Site Infections After Open Abdominal Surgery?
Brief Title: Clinical Outcome in View of Surgical Site Infection (SSI) With Antibacterial Skin Sutures
Status: Terminated | Type: Observational
Why Stopped: insufficient enrollment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: University Hospital Basel
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Wound Infection, Surgical
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort one with abdominal wall closure with Monocryl
- Cohort two with abdominal wall closure with Monocryl plus

SUMMARY:
Background: Poor wound healing and the development of surgical site infection (SSI) continue to occur and remain a significant cause of disability among operated patients. In spite of the substantial advances in our understanding of the epidemiology, pathogenesis and prevention it remains one of the most common complications in conventional abdominal surgery with an incidence in the literature between 4% and 17%. As it is known that surgical sutures potentiate the development of wound infection the search for an ideal suture material, suitable for all purposes has been pursued by surgeons for decades.

Hypothesis: In line with in-vitro results the investigators hypothesize that the use of antibacterial skin sutures with triclosan poliglecaprone 25 reduces the rate of SSI after open abdominal surgery Methods: To prevent microbial colonization of suture material in operative wounds and therefore to prevent SSI, triclosan-coated poliglecaprone 25 suture materials with antibacterial activity will be tested against un-coated suture material for skin closure after open abdominal surgery of 200 patients. The study is planed as a single center, randomized controlled trial. After ethical approval the patients will be consecutively enrolled from 2011 to 2012 in the Department of Visceral Surgery, University Hospital Basel, Switzerland. The patients will be followed for 30 days (day 3,7 and 30) to detect and document wound complications. Wound complications will be classified according to Center for Disease Control and Prevention Standard guidelines. Data will be collected and the rate of SSI will be analysed in both groups.

Expected value of the proposed project: If the investigators can confirm the proposed hypothesis in our study this could be a promising and feasible approach to lower SSI after open abdominal surgery and might be also used in other surgical fields. By lowering the rate of SSI the investigators might offer a new and cost saving procedure to the surgical community.

ELIGIBILITY:
Inclusion Criteria:

* All patients from the Visceral Department of Basel University Hospital requiring open abdominal surgery. Open abdominal surgery is defined as: opened peritoneal cavity

Exclusion Criteria:

* factors limiting the ability to co-operate in the study;
* absence of signed informed consent before entering the study;
* people with mental disorders;
* pregnant women;
* participants under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with required open abdominal surgery will be consecutively enrolled.Data of emergency patients are recorded separately as well as patients with a contaminated or dirty-infected (class III-IV) operative wound classified according to CDC guidelines on surgical wound classification1 further Patients with implanted foreign material such as mesh or vascular prosthesis.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Misteli, MD, Study Chair — Surgical Department of University Hospital Basel, Switzerland
Locations (1):
- Surgical Department of University Hospital Basel, Switzerland, Basel, Canton of Basel-City, Switzerland